CLINICAL TRIAL: NCT03158948
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 3 Doses of MOTREM in Patients With Septic Shock. A Randomised, Double-blind, Two-Stage, Placebo Controlled Study
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 3 Doses of MOTREM (Nangibotide) in Patients With Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inotrem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOT-C-201
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Shock, Septic
Keywords: Sepsis; LR12; TREM1; TREM-1
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — nangibotide

STUDY DESIGN:
Intervention Model Description: Randomised, Double-blind, Two-Stage, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- nangibotide 0.3 mg/kg/h (Experimental)
  Interventions: Drug: Nangibotide 0.3 mg/kg
- nangibotide 1.0 mg/kg/h (Experimental)
  Interventions: Drug: Nangibotide 1 mg/kg
- nangibotide 3.0 mg/kg/h (Experimental)
  Interventions: Drug: Nangibotide 3 mg/kg
- Placebo to nangibotide (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nangibotide 0.3 mg/kg — Formulated LR12 peptide
  Other Names: MOTREM 0.3 mg/kg
  Arms: nangibotide 0.3 mg/kg/h
Drug: Placebo — placebo
  Arms: Placebo to nangibotide
Drug: Nangibotide 1 mg/kg — Formulated LR12 peptide
  Other Names: MOTREM 1 mg/kg
  Arms: nangibotide 1.0 mg/kg/h
Drug: Nangibotide 3 mg/kg — Formulated LR12 peptide
  Other Names: MOTREM 3 mg/kg
  Arms: nangibotide 3.0 mg/kg/h

SUMMARY:
This is a randomised, double-blind, two-stage, placebo controlled study. It is designed to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of 3 doses of nangibotide versus placebo in adult patients with septic shock.

DETAILED DESCRIPTION:
This was a randomised, double-blind, two-stage, placebo-controlled study. It was composed of 2 stages with a similar treatment regimen in which 0.3, 1.0 or 3.0 mg/kg/h of nangibotide was tested versus placebo.

Stage 1 was performed to investigate ascending doses of nangibotide or placebo in a sequential design in cohorts of 4 patients (3:1 randomisation). After completion of a cohort (for up to 5 days of infusion), safety and available PK data were blindly reviewed by an independent data safety monitoring board (DSMB) before progressing to the next cohort. After completion of stage 1 DSMB evaluation, the study progressed to stage 2.

Stage 2 investigated 3 doses of nangibotide in a randomised, balanced, parallel-group design involving up to 3 doses of nangibotide and a placebo arm. Only dose arms of nangibotide considered to be safe and well tolerated during Stage 1 were to be administered in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent (proxy/legal representative) according to local regulations
* Age 18 to 80 years
* Documented or suspected infection: lung, abdominal or elderly UTI (≥65 years)
* Organ dysfunction defined as acute change in SOFA score ≥ 2 points
* Refractory hypotension requiring vasopressors to maintain MAP ≥65mm Hg despite adequate volume resuscitation of at least 20 ml/kg within 6 hours
* Hyperlactatemia (blood lactate >2 mmol/L or 18 mg/dL). This criterion must be met at least once for the purpose of diagnosis within the 24 hours before study drug administration

Exclusion Criteria: -

* Previous episode of septic shock (vasopressor administration) within current hospital stay
* Underlying concurrent immunodepression (specified in appendix 2)
* Solid organ transplant requiring immunosuppressive therapy
* Known pregnancy (positive serum pregnancy test)
* Prolonged QT syndrome (QTc ≥ 440 ms)
* Shock of any other cause, e.g. hypotension related to gastrointestinal bleeding
* Ongoing documented or suspected endocarditis, history of prosthetic heart valves
* End-stage neurological disease
* End-stage cirrhosis (Child Pugh Class C)
* Acute Physiology And Chronic Health Evaluation (APACHE) II score ≥ 34
* End stage chronic renal disease requiring chronic dialysis
* Home oxygen therapy on a regular basis for > 6 h/day
* Severe obesity (BMI ≥ 40)
* Recent CPR (within current hospital stay)
* Moribund patients
* Decision to limit full care taken before obtaining informed consent
* Participation in another interventional study in the 3 months prior to randomisation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno François, MD, Principal Investigator — Inserm 1435 Clinical Investigational Center, Limoges, France
Locations (4):
- Cliniques Universitaires Saint-Luc (there may be other sites in this country), Brussels, Belgium
- Inserm Clinical Investigational Center, CHU Dupuytren (there may be other sites in this country), Limoges, France
- Radboudumc (there may be other sites in this country), Nijmegen, Netherlands
- Hospital Clínico San Carlos, Medicina Intensiva (there may be other sites in this country), Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from 03 July 2017 (first patient first visit) to 11 June 2018 (last patient last visit) in 11 centers in 4 countries (Belgium, France, Spain, The Netherlands). 50 patients were included and randomized. 49 (98.0%) patients received the IMP and one patient died before IMP administration.
Pre-assignment Details: The duration of this study for each patient was a maximum of 13 weeks (including screening, up to 5 days of treatment and follow-up assessments 28 and 90 days after randomization). The purpose of the screening phase was to confirm patient eligibility for enrolment in the study based on the inclusion and exclusion criteria and to obtain written ICF.
Groups:
- Nangibotide 0.3 mg/kg/h: Nangibotide was administered as 5 mg/kg loading dose over 15 minutes followed by a continuous intravenous (i.v.) infusion at the dosage of 0.3 mg/kg/h for up to 5 days.
  MOTREM: 0.3 mg/kg/h Formulated LR12 peptide
- Nangibotide 1.0 mg/kg/h: Nangibotide was administered as 5 mg/kg loading dose over 15 minutes followed by a continuous intravenous (i.v.) infusion at the dosage of 1.0 mg/kg/h for up to 5 days.
  MOTREM: 1 mg/kg/hr Formulated LR12 peptide
- Nangibotide 3.0 mg/kg/h: Nangibotide was administered as 5 mg/kg loading dose over 15 minutes followed by a continuous intravenous (i.v.) infusion at the dosage of 3.0 mg/kg/h for up to 5 days.
  MOTREM: 3 mg/kg/h Formulated LR12 peptide
- Placebo: Placebo: placebo The matching placebo (solution of NaCl 0.9%) was administered as 5 mg/kg loading dose over 15 minutes followed by a continuous intravenous (i.v.) infusion at the dosage of 0.3 mg/kg/h for up to 5 days.
Period: Overall Study
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h | Placebo
Started | 13 | 12 | 12 | 12
Completed | 12 | 11 | 9 | 9
Not Completed | 1 | 1 | 3 | 3
Not completed — Death | 1 | 1 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Nangibotide 0.3 mg/kg/h: Nangibotide: 0.3 mg/kg Formulated LR12 peptide
- Nangibotide 1.0 mg/kg/h: Nangibotide: 1 mg/kg Formulated LR12 peptide
- Nangibotide 3.0 mg/kg/h: Nangibotide: 3 mg/kg Formulated LR12 peptide
- Total: Total of all reporting groups
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 12 | 12 | 49
Age, Customized [Count of Participants; unit: Participants]
  Age≤65 | 8 | 3 | 7 | 5 | 23
  Age>65 | 5 | 9 | 5 | 7 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 4 | 19
  Male | 7 | 7 | 8 | 8 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 13 | 9 | 11 | 8 | 41
  Black | 0 | 2 | 0 | 2 | 4
  Other | 0 | 1 | 1 | 2 | 4
Weight [Median (Full Range); unit: kg] | 75.0 [45 to 105] | 76.5 [45 to 108] | 68.0 [54 to 83] | 77.0 [42 to 99] | 74.0 [42 to 108]
Height [Median (Full Range); unit: cm] | 168.0 [155 to 186] | 168.5 [152 to 185] | 165.0 [150 to 185] | 167.5 [147 to 184] | 167.0 [147 to 186]
BMI [Median (Full Range); unit: kg/m^2] | 24.8 [17.1 to 37.2] | 26.0 [16.1 to 34.8] | 25.1 [18.1 to 36.8] | 27.5 [14.8 to 35.5] | 26.1 [14.8 to 37.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Treatment Emergent Adverse Events From Screening Until Study Completion
Description: Analyses were performed in the Safety Set composed of all randomized patients who received at least any dose of the study drug (nangibotide or placebo).
  Adverse events: Summary statistics of treatment emergent adverse events (TEAEs).
  Clinical events, including death, related to severe sepsis and sepsis complications were exempt from SAE reporting, unless the investigator deemed the event to be related to the administration of the study drug.
Time Frame: Adverse events experienced until D28 (End of study visit)
Population: Out of 49 patients included in all 4 groups, TEAEs were observed for 45 patients (12 patients experienced TEAEs in MOTREM 1 group, 12 patients experienced TEAEs in MOTREM 2 group, 11 patients experienced TEAEs in MOTREM 3 group and 10 patients experienced TEAEs in placebo group)
Measure: Count of Participants; unit: Participants
Groups:
- Nangibotide 0.3 mg/kg/h; Nangibotide 1.0 mg/kg/h; Nangibotide 3.0 mg/kg/h: Nangibotide: Formulated LR12 peptide
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h | Placebo
Number analyzed (Participants) | 13 | 12 | 12 | 12
Participants | 12 | 12 | 11 | 10

2. Primary Outcome: Systolic Blood Pressure (SBP)
Description: Systolic blood pressure measured by sphygmomanometer at study site. Median SBP at each visit is summarized by treatment group.
Time Frame: Vital signs were assessed each day from day zero (D0 [before investigational medicinal product initiation]) to end of infusion at day 5 (D5) and on final study day at day 28 (D28).
Population: The data is not available for all subjects and the data in the tables below refers to only those participants who were measured and analyzed. Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), Mean Arterial Pressure (mmHg), heart rate (bpm) and temperature in Celsius degrees were described at each time when it was available: D1, D2, D3, D4, D5 and EOS visit.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
mmHg
  D0: number analyzed (Participants) | 10 | 13 | 12 | 12
  D0 | 121.5 [87 to 149] | 110.0 [90 to 133] | 121.0 [96 to 131] | 111.0 [87 to 160]
  D1: number analyzed (Participants) | 8 | 9 | 10 | 11
  D1 | 114.5 [82 to 131] | 117.0 [96 to 159] | 112.5 [93 to 124] | 113.0 [97 to 150]
  D2: number analyzed (Participants) | 2 | 4 | 5 | 7
  D2 | 107.0 [104 to 110] | 116.0 [96 to 147] | 121.0 [105 to 130] | 112.0 [100 to 150]
  D3: number analyzed (Participants) | 2 | 2 | 4 | 4
  D3 | 94.0 [87 to 101] | 126.5 [124 to 129] | 108.5 [96 to 127] | 112.5 [102 to 123]
  D4: number analyzed (Participants) | 2 | 1 | 3 | 4
  D4 | 108.0 [104 to 112] | 133.0 [133 to 133] | 105.0 [101 to 125] | 107.0 [95 to 119]
  D5/EOI: number analyzed (Participants) | 10 | 13 | 12 | 12
  D5/EOI | 117.0 [80 to 137] | 118.0 [94 to 180] | 114.5 [99 to 170] | 109.0 [79 to 131]
  D28/EOS: number analyzed (Participants) | 9 | 11 | 11 | 9
  D28/EOS | 135.0 [107 to 181] | 120.0 [90 to 140] | 111.0 [95 to 166] | 113.0 [93 to 120]

3. Primary Outcome: Diastolic Blood Pressure (DBP)
Description: Median DBP at each visit is summarized by treatment group.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: mmHg
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
mmHg
  D0: number analyzed (Participants) | 10 | 13 | 12 | 12
  D0 | 53.5 [44 to 77] | 55.0 [40 to 78] | 59.0 [49 to 78] | 55.5 [44 to 72]
  D1: number analyzed (Participants) | 8 | 9 | 10 | 11
  D1 | 59.0 [45 to 72] | 55.0 [32 to 75] | 59.5 [48 to 128] | 58.0 [44 to 75]
  D2: number analyzed (Participants) | 2 | 4 | 5 | 7
  D2 | 61.0 [56 to 66] | 63.5 [61 to 75] | 66.0 [58 to 72] | 67.0 [47 to 86]
  D3: number analyzed (Participants) | 2 | 2 | 4 | 4
  D3 | 58.5 [50 to 67] | 60.5 [60 to 61] | 55.5 [40 to 62] | 62.0 [46 to 70]
  D4: number analyzed (Participants) | 2 | 1 | 3 | 4
  D4 | 61.5 [55 to 68] | 64.0 [64 to 64] | 55.0 [52 to 56] | 58.0 [46 to 63]
  D5/EOI: number analyzed (Participants) | 10 | 13 | 12 | 12
  D5/EOI | 55.5 [46 to 63] | 58.0 [38 to 95] | 57.0 [44 to 81] | 57.0 [30 to 71]
  D28/EOS: number analyzed (Participants) | 9 | 11 | 11 | 9
  D28/EOS | 70.0 [40 to 82] | 70.0 [35 to 90] | 60.0 [45 to 80] | 65.0 [60 to 80]

4. Primary Outcome: Median Arterial Pressure (MAP)
Description: MAP at each visit is summarized by treatment group.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: mmHg
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
mmHg
  D0: number analyzed (Participants) | 10 | 13 | 12 | 12
  D0 | 72.0 [61 to 101] | 71.0 [60 to 98] | 78.0 [67 to 96] | 73.0 [61 to 116]
  D1: number analyzed (Participants) | 8 | 9 | 10 | 11
  D1 | 77.5 [57 to 92] | 76.0 [60 to 97] | 74.0 [55 to 87] | 77.0 [65 to 100]
  D2: number analyzed (Participants) | 2 | 4 | 5 | 7
  D2 | 76.0 [69 to 83] | 82.5 [77 to 105] | 80.0 [55 to 90] | 80.0 [67 to 98]
  D3: number analyzed (Participants) | 2 | 2 | 4 | 4
  D3 | 71.0 [62 to 80] | 84.5 [84 to 85] | 72.5 [54 to 83] | 79.0 [70 to 88]
  D4: number analyzed (Participants) | 2 | 1 | 3 | 4
  D4 | 76.5 [69 to 84] | 92.0 [92 to 92] | 71.0 [69 to 74] | 77.0 [70 to 79]
  D5/EOI: number analyzed (Participants) | 10 | 13 | 12 | 12
  D5/EOI | 75.0 [58 to 82] | 78.0 [61 to 130] | 76.0 [59 to 112] | 72.5 [41 to 90]
  D28/EOS: number analyzed (Participants) | 8 | 10 | 11 | 9
  D28/EOS | 87.0 [62 to 99] | 86.5 [52 to 106] | 74.0 [59 to 107] | 79.0 [66 to 93]

5. Primary Outcome: Heart Rate
Description: Median heart rate at each visit is summarized by treatment group.
Time Frame: Vital signs were assessed each day from day zero (D0 [before investigational medicinal product initiation]) to end of infusion at day 5 (D5).
Population: The data is not available for all subjects and the data in the tables below refers to only those participants who were measured and analyzed. systolic blood pressure (mmHg). Diastolic blood pressure (mmHg), mean arterial pressure (mmHg), heart rate (bpm) and temperature i celcius degrees were described at each time when it was available: D0, D1, D2, D3, D4 and D5/EOI visit.
Measure: Median (Full Range); unit: bpm
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
bpm
  D0: number analyzed (Participants) | 10 | 13 | 12 | 12
  D0 | 83.5 [54 to 136] | 94.0 [75 to 138] | 104.5 [66 to 136] | 97.5 [85 to 147]
  D1: number analyzed (Participants) | 8 | 9 | 10 | 11
  D1 | 89.0 [58 to 145] | 86.0 [70 to 135] | 91.0 [65 to 131] | 98.0 [77 to 135]
  D2: number analyzed (Participants) | 2 | 4 | 5 | 7
  D2 | 74.0 [60 to 88] | 85.0 [80 to 105] | 110.0 [92 to 132] | 83.0 [58 to 153]
  D3: number analyzed (Participants) | 2 | 2 | 4 | 4
  D3 | 95.0 [70 to 120] | 60.5 [58 to 63] | 102.5 [61 to 121] | 88.5 [64 to 100]
  D4: number analyzed (Participants) | 2 | 1 | 3 | 4
  D4 | 75.0 [70 to 80] | 61.0 [61 to 61] | 121.0 [100 to 156] | 84.5 [66 to 96]
  D5/EOI: number analyzed (Participants) | 10 | 13 | 12 | 12
  D5/EOI | 86.0 [67 to 129] | 91.0 [55 to 133] | 93.5 [58 to 112] | 91.0 [70 to 122]

6. Primary Outcome: Temperature
Description: Median temperature at each visit is summarized by treatment group.
Time Frame: as for outcome 5
Population: The data is not available for all subjects and the data in the tables below refers to only those participants who were measured and analyzed. Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), Mean Arterial Pressure (mmHg), heart rate (bpm) and temperature in Celsius degrees were described at each time when it was available: D0, D1, D2, D3, D4, D5/EOI visit.
Measure: Median (Full Range); unit: °C
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
°C
  D0: number analyzed (Participants) | 10 | 13 | 12 | 12
  D0 | 37.3 [35 to 38.9] | 36.8 [35.7 to 38.9] | 37.0 [35.8 to 38.5] | 37.0 [34 to 39.6]
  D1: number analyzed (Participants) | 8 | 9 | 10 | 11
  D1 | 36.3 [35.5 to 40.8] | 36.2 [33.5 to 39.3] | 36.8 [36 to 38] | 37.1 [35.7 to 38.8]
  D2: number analyzed (Participants) | 2 | 4 | 5 | 7
  D2 | 36.1 [35.5 to 36.6] | 36.3 [35.7 to 37] | 36.5 [36 to 37.4] | 37.4 [35.1 to 38.9]
  D3: number analyzed (Participants) | 2 | 2 | 4 | 4
  D3 | 36.6 [36 to 37.1] | 36.3 [35.6 to 36.9] | 36.7 [36.1 to 37.8] | 37.4 [36.1 to 38.2]
  D4: number analyzed (Participants) | 2 | 1 | 3 | 4
  D4 | 36.1 [36 to 36.2] | 36.1 [36.1 to 36.1] | 36.9 [36.6 to 37.4] | 36.6 [36.3 to 37.3]
  D5/EOI: number analyzed (Participants) | 10 | 13 | 12 | 12
  D5/EOI | 36.9 [35.8 to 37.3] | 36.2 [35.6 to 37.9] | 36.5 [35.4 to 38.6] | 36.4 [34.3 to 38.3]

7. Primary Outcome: Electrocardiogram
Description: Abnormal and emergent clinically significant electrocardiogram were summarized for each group.
Time Frame: Electrocardiogram was performed each day from D0 (before IMP initiation) to D5 (EOI) and on D28 (EOS).
Population: Some patients did not perform ECG at some visits
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
Participants
  ECG - D1: number analyzed (Participants) | 12 | 9 | 9 | 12
  ECG - D1: ECGs - Normal | 4 | 1 | 4 | 5
  ECG - D1: ECGs - Abnormal NCS | 3 | 4 | 4 | 5
  ECG - D1: ECGs - Abnormal CS | 5 | 4 | 1 | 2
  ECG - D1: ECGs - Missing | 0 | 0 | 0 | 0
  ECG - D2: number analyzed (Participants) | 2 | 4 | 5 | 6
  ECG - D2: ECGs - Normal | 1 | 2 | 1 | 4
  ECG - D2: ECGs - Abnormal NCS | 0 | 1 | 2 | 0
  ECG - D2: ECGs - Abnormal CS | 1 | 1 | 2 | 2
  ECG - D2: ECGs - Missing | 0 | 0 | 0 | 0
  ECG - D3: number analyzed (Participants) | 2 | 2 | 3 | 4
  ECG - D3: ECGs - Normal | 0 | 1 | 0 | 2
  ECG - D3: ECGs - Abnormal NCS | 1 | 1 | 2 | 1
  ECG - D3: ECGs - Abnormal CS | 1 | 0 | 1 | 1
  ECG - D3: ECGs - Missing | 0 | 0 | 0 | 0
  ECG - D4: number analyzed (Participants) | 1 | 1 | 3 | 4
  ECG - D4: ECGs - Normal | 0 | 1 | 0 | 2
  ECG - D4: ECGs - Abnormal NCS | 1 | 0 | 1 | 1
  ECG - D4: ECGs - Abnormal CS | 0 | 0 | 2 | 1
  ECG - D4: ECGs - Missing | 0 | 0 | 0 | 0
  ECG - D5/EOI: number analyzed (Participants) | 9 | 11 | 8 | 12
  ECG - D5/EOI: ECGs - Normal | 3 | 3 | 4 | 4
  ECG - D5/EOI: ECGs - Abnormal NCS | 4 | 7 | 3 | 4
  ECG - D5/EOI: ECGs - Abnormal CS | 2 | 1 | 1 | 4
  ECG - D5/EOI: ECGs - Missing | 0 | 0 | 0 | 0
  ECG - D28/EOS: number analyzed (Participants) | 9 | 8 | 11 | 9
  ECG - D28/EOS: ECGs - Normal | 3 | 5 | 4 | 4
  ECG - D28/EOS: ECGs - Abnormal NCS | 5 | 3 | 6 | 4
  ECG - D28/EOS: ECGs - Abnormal CS | 1 | 0 | 1 | 1
  ECG - D28/EOS: ECGs - Missing | 0 | 0 | 0 | 0

8. Primary Outcome: Anti-Drug Antibodies (ADA Dimer)
Description: Anti-Drug Antibodies test was performed for all patients.
Time Frame: Anti-Drug Antibodies test were done at D0, D10 and D28 in all patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
Participants
  D0: MISSING | 0 | 0 | 0 | 0
  D0: NEGATIVE | 12 | 13 | 12 | 12
  D0: POSITIVE | 0 | 0 | 0 | 0
  D10: MISSING | 11 | 13 | 9 | 7
  D10: NEGATIVE | 1 | 0 | 3 | 5
  D10: POSITIVE | 0 | 0 | 0 | 0
  D28: MISSING | 3 | 4 | 2 | 3
  D28: NEGATIVE | 9 | 9 | 10 | 9
  D28: POSITIVE | 0 | 0 | 0 | 0

9. Primary Outcome: Anti-Drug Antibodies (ADA Monomer)
Description: Anti-Drug Antibodies test was performed for all patients.
Time Frame: Anti-Drug Antibodies test were measured at D0, D10 and D28.
Population: The results are presented for the Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 12 | 13 | 12 | 12
Participants
  D0: MISSING | 0 | 0 | 0 | 0
  D0: NEGATIVE | 12 | 13 | 12 | 12
  D0: POSITIVE | 0 | 0 | 0 | 0
  D10: MISSING | 11 | 13 | 9 | 7
  D10: NEGATIVE | 1 | 0 | 3 | 5
  D10: POSITIVE | 0 | 0 | 0 | 0
  D28: MISSING | 3 | 5 | 2 | 3
  D28: NEGATIVE | 9 | 8 | 10 | 9
  D28: POSITIVE | 0 | 0 | 0 | 0

10. Secondary Outcome: Pharmacokinetic Parameters From the Non-compartmental Analysis: Cmax
Description: As no pharmacokinetic sample was planned just after the loading dose, maximum observed nangibotide plasma concentration (Cmax) was in the same magnitude as steady-state concentration during the maintenance infusion, calculated as the median of the observed pre-dose concentration from day2 onwards up to the last pre-dose concentration available in the study (Cavg).
Time Frame: Baseline: pre-dose sample at Day 0 (D0) Daily up to Day 5 (D5) (or the last day in the study/EOI) If possible, at D5/EOI: - 15 min before end of infusion (EOI) - 10 min after EOI - 30 min after EOI - 2h after EOI
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 13 | 12 | 12
ng/mL | 71.2 [20.0 to 219] | 234 [71.3 to 514] | 914 [502 to 6095]

11. Secondary Outcome: Pharmacokinetic Parameters From the Non-compartmental Analysis: Tmax
Description: Time to reach the maximum observed nangibotide plasma concentration (h) was measured for all groups.
Time Frame: as for outcome 10
Measure: Median (Full Range); unit: h
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 13 | 12 | 12
h | 22.7 [14.3 to 76.0] | 25.4 [9.25 to 118] | 36.0 [9.00 to 75.8]

12. Secondary Outcome: Pharmacokinetic Parameters From the Non-compartmental Analysis: AUC0-last
Description: Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration Clast was calculated using the log-linear trapezoidal method.
Time Frame: as for outcome 10
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 13 | 12 | 12
ng*h/mL | 1722 [360 to 5243] | 7579 [668 to 45189] | 47320 [3830 to 393506]

13. Secondary Outcome: Pharmacokinetic Parameters From the Non-compartmental Analysis: Cavg
Description: Steady-state concentration during the maintenance infusion was calculated as the median of the observed pre-dose concentration from day2 onwards up to the last pre-dose concentration available in the study.
Time Frame: as for outcome 10
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 13 | 12 | 12
ng/mL | 67.6 [20.0 to 219] | 223 [71.3 to 418] | 729 [93.9 to 3778]

14. Secondary Outcome: Pharmacokinetic Parameters From the Non-compartmental Analysis: CL
Description: Systemic clearance was calculated as the ratio between the infusion rate during the maintenance infusion and Cavg.
Time Frame: as for outcome 10
Measure: Median (Full Range); unit: L/h/kg
Arm/Group | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
Number analyzed (Participants) | 13 | 12 | 12
L/h/kg | 4.52 [1.36 to 15.3] | 4.50 [2.39 to 14.0] | 4.12 [0.794 to 25.0]

ADVERSE EVENTS:
Time Frame: From baseline until D28
Description: All deaths, Serious Adverse Events, and Other Adverse Events are reported in the Adverse Event module.
Groups:
- Nangibotide 0.3 mg/kg/h; Nangibotide 1.0 mg/kg/h; Nangibotide 3.0 mg/kg/h: MOTREM: Formulated LR12 peptide
Arm/Group | Placebo | Nangibotide 0.3 mg/kg/h | Nangibotide 1.0 mg/kg/h | Nangibotide 3.0 mg/kg/h
All-Cause Mortality (participants affected / at risk) | 3/12 | 4/13 | 2/12 | 4/12
Serious Adverse Events (participants affected / at risk) | 7/12 | 4/13 | 2/12 | 4/12
Other Adverse Events (participants affected / at risk) | 10/12 | 12/13 | 12/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Nangibotide 0.3 mg/kg/h (N=13) | Nangibotide 1.0 mg/kg/h (N=12) | Nangibotide 3.0 mg/kg/h (N=12)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ failure syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Nangibotide 0.3 mg/kg/h (N=13) | Nangibotide 1.0 mg/kg/h (N=12) | Nangibotide 3.0 mg/kg/h (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (5) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Confusional State (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Intra-Abdominal Fluid Collection (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT03158948/Prot_SAP_000.pdf